CLINICAL TRIAL: NCT02371603
Title: An Open Label, Randomized, Two Part Study to Evaluate the CYP2C8- and OATP1B1-Mediated Drug-Drug Interaction Potential of GSK1278863 With Pioglitazone and Rosuvastatin as Victims and Trimethoprim as Perpetrator in Healthy Adult Volunteers
Brief Title: Drug-drug Interaction Study of GSK1278863 With Pioglitazone, Rosuvastatin and Trimethoprim in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200229
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Anaemia
Keywords: Prolyl hydroxylase inhibitor; GSK1278863; Anemia; Drug interaction
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Tablets; Pioglitazone; Rosuvastatin Calcium; Trimethoprim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: GSK1278863, pioglitazone and rosuvastatin (Experimental): Subjects will receive single, oral 15 milligram (mg) pioglitazone, 10 mg rosuvastatin and 25 mg dose of GSK1278863 (Treatment A) or 15 mg pioglitazone and 10 mg rosuvastatin (Treatment B) on Day 1 and a 25 mg dose of GSK1278863 alone on Day 2 in two treatment periods as per treatment sequence AB or BA. The 2 treatment periods will be separated by a wash out period of approximately 7 days
  Interventions: Drug: GSK1278863 25 mg Tablet; Drug: Pioglitazone 15 mg Tablet; Drug: Rosuvastatin 10 mg Tablet
- Part B: GSK1278863 and trimethoprim (Experimental): Subjects will receive a single, oral 25 mg dose of GSK1278863 on Day 1 and Day 6 morning. The subjects will also receive 200 mg dose of trimethoprim twice daily from Day 3 to 6, with Day 6 dosing being concomitant with morning dosing of GSK1278863
  Interventions: Drug: GSK1278863 25 mg Tablet; Drug: Trimethoprim 100 mg Tablet

INTERVENTIONS:
Drug: GSK1278863 25 mg Tablet — A round, biconvex, white film coated tablet to be taken orally in the fasted state in the morning
Drug: Pioglitazone 15 mg Tablet — White to off-white, round, convex, non scored tablet with "ACTOS" on one side, and "15" on the other, to be taken orally in the fasted state in the morning
  Arms: Part A: GSK1278863, pioglitazone and rosuvastatin
Drug: Rosuvastatin 10 mg Tablet — Pink, round, biconvex, coated tablets. Debossed "CRESTOR" and "10" on one side, to be taken orally in the fasted state in the morning
  Arms: Part A: GSK1278863, pioglitazone and rosuvastatin
Drug: Trimethoprim 100 mg Tablet — White, round, scored, convex tablet, debossed "93" above the score and debossed "2159" below the score on one side and plain on the other, to be taken orally as two tablets once in the morning and once in the evening
  Arms: Part B: GSK1278863 and trimethoprim

SUMMARY:
This study will be a two-part with an open-label, single oral dose, two-way crossover study design. Part A and Part B of the study are independent and may be conducted in parallel. The Part A of the study will assess the effect of an oral dose of GSK1278863 on the pharmacokinetics of a CYP2C8 (pioglitazone) and OATP1B1 (rosuvastatin) probe substrate in order to determine the potential for clinically-significant drug interactions with CYP2C8 and OATP1B1 substrates. The Part B of the study will assess the effect of a weak CYP2C8 inhibitor (trimethoprim) on the pharmacokinetics of GSK1278863 and its six predominant metabolites. Part A will be conducted in approximately 30 healthy subjects, having a randomized study design. There will be approximate 7-day washout period between each dosing period. Part B will be conducted in approximately 20 healthy subjects, having single sequence study design. Follow up will be conducted within 7 to 10 days after the last dose in both Part A and B. The total duration of a subject's involvement in the part A of the study will be approximately 8 weeks (Screening to Follow-up) and in part B will be approximately 7 weeks (Screening to Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 18 and 65 years of age, inclusive at the time of signing the informed consent form.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and ECG monitoring obtained at the screening visit. The determination of clinical significance will be made by the investigator and the GlaxoSmithKline (GSK) Medical Monitor and will require that the finding is unlikely to introduce additional risk factors or interfere with the study procedures, or the integrity of the study.
* Hemoglobin values at screening greater than the lower limit of the laboratory reference range and less than or equal to 16.0 grams (g)/ deciliter (dL) for males and less than or equal to 14.0 g/dL for females.
* Body weight >=50 Kilogram (kg) and Body Mass Index (BMI) within the range 19-29.9 kg/meter (m)^2 (inclusive).
* Female or Male. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine or serum human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: a) Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation and Documented hysteroscopic tubal occlusion procedure with follow-up, confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy, b) Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) 23.0-116.3 International units (IU)/ liter (L) and estradiol levels consistent with menopause (<32 picogram (pg)/ milliliter [mL]) are confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrolment. c) Reproductive potential and agrees to follow the contraception requirement for Female Subjects from 30 days prior to the first dose of study treatment and until at least five terminal half-lives or until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study treatment and completion of the follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine transaminase (ALT), alkaline phosphatase and bilirubin >1.5xUpper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT interval(QTc): QT interval corrected for heart rate according to Bazetts formula (QTcB) >450 milliseconds (msec), The QTc must be the QT interval corrected for heart rate according to Bazetts formula (QTcB). For purposes of data analysis, QTcB will be used.
* Hypertensive (diastolic Blood pressure (BP) >90 millimetre of mercury (mmHg) or systolic BP >140 mmHg at Screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of deep vein thrombosis, stroke, transient ischemic attack, pulmonary embolism or other thrombosis related condition.
* History of myocardial infarction or acute coronary syndrome.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of GSK1278863, trimethoprim, pioglitazone or rosuvastatin. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue.
* Evidence of active peptic, duodenal or esophageal ulcer disease at Screening or history of clinically significant Gastrointestine (GI) bleeding.
* Subjects with chronic inflammatory joint disease (example [e.g.]., scleroderma, systemic lupus erythematosis, rheumatoid arthritis).
* Subjects with a history of pulmonary artery hypertension.
* Subjects with a history of malignancy within the prior five years, who are receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders); with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to screening through Day -1 (Randomization).
* History of proliferative vascular eye disease (e.g., choroidal or retinal disease, such as neovascular age-related macular degeneration, proliferative diabetic retinopathy or macular edema).
* Subjects with heart failure, as defined by the New York Heart Association (NYHA) functional classification system, including known right heart failure
* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) except occasional usage of acetaminophen, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the follow-up visit, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products prior to screening.
* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to any of the study treatments (e.g., GSK1278863, pioglitazone, rosuvastatin, trimethoprim), or their components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Consumption of >3 servings/day of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of investigational product until the follow-up visit, unless in the opinion of the investigator and GSK Medical Monitor this will not interfere with the study procedures or compromise subject safety.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the study treatment (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2015-08-12 (Actual); Study Completion 2015-08-12 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters for pioglitazone following oral administration of pioglitazone alone and in combination with GSK1278863, evaluated by measurement of plasma Cmax and AUC (0-infinity) for Part A | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours (h) post-dose in each treatment period
  The effect of an oral dose of GSK1278863 on the pharmacokinetics of pioglitazone will be assessed using the following PK parameters: maximum observed concentration (Cmax), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC (0-infinity)
Composite of PK parameters for rosuvastatin following oral administration of rosuvastatin alone and in combination with GSK1278863 evaluated by measurement of plasma Cmax and AUC (0-infinity) for Part A | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 h post-dose in each treatment period
  The effect of an oral dose of GSK1278863 on the pharmacokinetics of rosuvastatin will be assessed using the following PK parameters: Cmax and AUC (0-infinity)
Composite of PK parameters for GSK1278863 and its 6 predominant metabolites following oral administration of GSK1278863 alone and in combination with steady-state trimethoprim evaluated by measurement of plasma Cmax and AUC (0-infinity) for Part B | Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, and 48 h post-dose of GSK1278863 on day 1 and day 6
  The effect of trimethoprim on the pharmacokinetics of GSK1278863 and six predominant metabolites (GSK2391220 [M2], GSK2506104 [M3], GSK2487818 [M4], GSK2506102 [M5], GSK2531398 [M6], GSK2531401 [M13]) will be assessed using the following PK parameters: Cmax and AUC (0-infinity)

SECONDARY OUTCOMES:
Composite of PK parameters for pioglitazone following oral administration of pioglitazone alone and in combination with GSK1278863 evaluated by measurement of plasma AUC(0-t), tmax and t1/2 for Part A | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 h post-dose in each treatment period
  Additional plasma PK parameters for characterizing the effect of co-administration of GSK1278863 on the pharmacokinetics of pioglitazone are the following: area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC[0-t]), time of occurrence of Cmax (tmax) and terminal phase half-life (t1/2)
Composite of PK parameters for rosuvastatin following oral administration of rosuvastatin alone and in combination with GSK1278863 evaluated by measurement of plasma AUC(0-t), tmax and t1/2 for Part A | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 h post-dose in each treatment period
  Additional plasma PK parameters for characterizing the effect of co-administration of GSK1278863 on the pharmacokinetics of rosuvastatin are the following: AUC[0-t], tmax) and t1/2
Composite of PK parameters for GSK1278863 and its 6 predominant metabolites following oral administration ofGSK1278863 alone and in combination withsteady-state trimethoprim evaluated by measurement of plasma AUC(0-t), tmax and t1/2 for Part B | Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, and 48 h post-dose of GSK1278863 on day 1 and day 6
  Additional plasma PK parameters for characterizing the effect of co-administration of steady-state trimethoprim on the pharmacokinetics of GSK1278863 and six predominant metabolites (GSK2391220 [M2], GSK2506104 [M3], GSK2487818 [M4],GSK2506102 [M5], GSK2531398 [M6],GSK2531401 [M13]) are the following: AUC[0-ttmax and t1/2
Number of participants with adverse events as a measure of safety and tolerability of GSK1278863 alone and co-administered with pioglitazone and rosuvastatin or steady-state trimethoprim | Up to 4 weeks for Part A and up to 3 weeks for Part B
  Adverse events will be collected from Day -1 and until the final follow-up visit. Intensity of AEs will be categorized as mild, moderate or severe
Composite of clinical laboratory tests assessed by measuring hematology, clinical chemistry and urinalysis | Up to 4 weeks for Part A and up to 3 weeks for Part B
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis
Safety and tolerability of single oral dose of GSK1278863 alone and co-administered with pioglitazone and rosuvastatin or steady-state trimethoprim assessed by12-lead electrocardiogram (ECG) | Up to 4 weeks for Part A and up to 3 weeks for Part B
  Triplicate 12-lead ECGs will be obtained at each timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals
Composite of vital signs assessed by measuring temperature, systolic and diastolic blood pressure and pulse rate | Up to 4 weeks for Part A and up to 3 weeks for Part B
  Vital signs will be measured in supine position after 5 minutes rest and will include temperature, systolic and diastolic blood pressure and pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200229 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200229?search=study&b'study_ids=200229'#rs
- Available data/document: Informed Consent Form: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200229 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register